CLINICAL TRIAL: NCT03367169
Title: Comparison of the Minimally Invasive Surgery Versus Open Reduction in the Surgery of the Pilon Fractures
Brief Title: Surgery of the Pilon Fractures
Acronym: MICOPIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recrutment problems
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-368; 2017-A01735-48 (Other: 2017-A01735-48)
Record Dates: First submitted 2017-11-23; First posted 2017-12-08 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Pilon Fractures; Fractures; Bone; Leg Injuries
Keywords: Pilon fractures; Osteosynthesis; Mini invasive plate osteosynthesis; Locked plate; Open reduction
MeSH Terms: conditions — Fractures, Bone; Leg Injuries

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive method (Active Comparator): The patients are treated with minimally invasive method
  Interventions: Procedure: minimally invasive method
- open reduction method (Active Comparator): The patients are treated with open reduction method
  Interventions: Procedure: open reduction method

INTERVENTIONS:
Procedure: minimally invasive method — type of surgical technique
  Arms: minimally invasive method
Procedure: open reduction method — type of surgical technique
  Arms: open reduction method

SUMMARY:
The assessment consists in comparing the osteosynthesis plate with minimally invasive technique versus open reduction and internal fixation.

The aim of study is to compare (period of bandage, efficacy, safety), these two types of surgical technique by using a prospective, randomized analysis.

DETAILED DESCRIPTION:
Several surgical techniques exist and among plate osteosynthesis, there is a minimally invasive method and the open reduction method.

Investigators think that the minimally invasive method with intern plate is more efficient than the open reduction method.

These techniques may better preserve perifracture soft tissues, hematoma. It may lead to a smaller muscle detachment.

The minimally invasive technique allows a more efficient vascularization of the fracture site, what would increase bone healing and the functional prognosis of tibial pilon lesions.

It's all these issues investigators would like to assess with a randomized study.

ELIGIBILITY:
Inclusion Criteria:

* More than 18-year-old with opened or closed pilon fracture Cauchoix type 1,
* signed patient consent

Exclusion Criteria:

* Open pilon fracture cauchoix type 2 or 3,
* infection of the operating site,
* previous osseous disease
* patient who are unwilling or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Healing | at 45 days
  Measure of the duration of the bandage with index form of follow-up the state cutaneous of the wound. This measure was a number.

SECONDARY OUTCOMES:
AOFAS clinical score | pre op, 45 days, 3, 6 and 12 months
  American Orthopedic Foot and Ankle Society was a standard method of reporting clinical status of the ankle and foot. The systems incorporate both subjective and objective factors into numerical scales to describe function, alignment, and pain. The score varies between 0 and 100, more the value is better brought up is the score
Nach mazur and al score | pre op 45 days, 3, 6 and 12 months
  The Nach mazur grading system uses 100 points to assess pain, function while wearing shoes and the range of ankle movement. The maximum score a patient with a solid ankle fusion.
The Foot & Ankle Disability Index | pre op 45 days, 3, 6 and 12 months
  The Foot and Ankle Disability Index (FADI) was designed to assess functional limitations related to foot and ankle conditions. Subjective reports of function are classified as generic or specific measures, which include condition-specific, population-specific, and patient-specific instruments. The FADI have a total point value of 100 points, more the value is better brought up is the score
Pain | pre op 45 days, 3, 6 and 12 months
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
Complications | pre op 45 days, 3, 6 and 12 months
  list of the complications
Radiologic evaluation | pre op 45 days, 3, 6 and 12 months
  Radiologic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Roger ERIVAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France